CLINICAL TRIAL: NCT02645279
Title: Comparison of Oral 30 % Dextrose and iv Midazolam Sedation During MRI in Neonates
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, H. Evren Eker, Ass Prof, Baskent University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: KA15/19
Record Dates: First submitted 2015-12-30; First posted 2016-01-01 (Estimated); Last update posted 2016-01-01 (Estimated); Status verified 2015-12

CONDITIONS: Epilepsy; Trauma; Metabolic Disease
Keywords: newborn; MRI; oral 30% glucose
MeSH Terms: conditions — Epilepsy; Wounds and Injuries; Metabolic Diseases | interventions — Glucose; Midazolam

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- oral 30% glucose (Active Comparator): oral 30% glucose total 200 mg/kg with 0.5-1 mL increments
  Interventions: Other: oral 30% glucose
- IV midazolam (Active Comparator): intravenous administration of midazolam 0.1 mg/kg
  Interventions: Drug: IV midazolam

INTERVENTIONS:
Other: oral 30% glucose — 30% glucose solution was administered orally through a teat. 1 mL 30% glucose solution was added following placement of the teat into the mouth of the newborn. After suckling of 0.5-1 mL glucose solution, the motionless and sleepiness of newborn was evaluated. If the target conditions was not achieved, 0.5-1 mL increments of glucose was added until the newborn kept motionless or asleep.
  Arms: oral 30% glucose
Drug: IV midazolam — IV 0.1 mg/kg midazolam was administered.MRI was routinely performed and the newborns who did not keep motionless or asleep and had motion artefacts were sedated with intravenous 0.5 mg/kg propofol.
  Arms: IV midazolam

SUMMARY:
The purpose of this study is to demonstrate the effectiveness of oral glucose administration during MRI for imaging of newborns and compare with midazolam sedation.

DETAILED DESCRIPTION:
Motion artefacts affect the quality of MRI and in order to overcome this problem procedures are performed under sedation or general anaesthesia. The safety profile of these methods for newborns is unclear. Alternative non-pharmacological interventions are changeable and might be time consuming. Oral glucose/sucrose administration has been the most frequently studied non-pharmacologic intervention in term and preterm neonates during painful procedures. In this study investigators aimed to compare oral 30% glucose and intravenous midazolam their efficiency on sedation during MRI.

ELIGIBILITY:
Inclusion Criteria:

* Neonates requiring MR imaging for diagnosis

Exclusion Criteria:

* Patients with fever, cold symptoms, suspicion of difficult airway, hypovolemia, cardiac, renal, lung disease, malformations

Ages: 1 Day to 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 112 (Actual)
Dates: Start 2015-01; Primary Completion 2016-02 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
Success rate of the procedures to keep the neonates quietened, motionless and slept during the procedure and to consider all images qualitatively appropriate for interpretation | Approximately 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Anis Aribogan, Prof, Study Chair — Baskent University Department of Anesthesiology